CLINICAL TRIAL: NCT00067626
Title: Chromium Effects on Insulin and Vascular Function in People at Risk for Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Yale University (Other)
Responsible Party: David L. Katz, MD, MPH, Yale-Griffin Prevention Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R21AT001332 (NIH); R21AT001332 (NIH)
Record Dates: First submitted 2003-08-25; First posted 2003-08-26 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Obesity; Pre-diabetes; Insulin Resistance; Impaired Glucose Tolerance; Impaired Fasting Glucose
Keywords: glucose tolerance test; minerals; chromium; complementary and alternative medicine
MeSH Terms: conditions — Obesity; Glucose Intolerance; Insulin Resistance | interventions — Chromium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 500/1000 mcg oral chromium taken daily or placebo (crossover)
  Interventions: Dietary Supplement: Chromium
- 2 (Experimental): 500/1000 mcg oral chromium taken daily or placebo (crossover)
  Interventions: Dietary Supplement: Chromium

INTERVENTIONS:
Dietary Supplement: Chromium — 500/1000 mcg oral chromium picolinate taken daily or placebo (crossover)

SUMMARY:
The purpose of this study is to investigate the effects of Chromium on glucose tolerance and endothelial function in people at risk for type II diabetes.

DETAILED DESCRIPTION:
Impaired glucose tolerance (IGT), impaired fasting glucose (IFG), and insulin resistance (IR) are precursors to type II diabetes mellitus (DM) and its sequelae, and are cardiac risk factors in their own right. The worsening epidemic of DM in the US, along with the increasing prevalence of obesity, insulin resistance, and IGT, render the identification of promising interventions for these states a matter of some urgency. While lifestyle interventions based on dietary pattern and physical activity can delay or prevent the onset of diabetes, and reduce cardiovascular risk, adherence at the population level is severely limiting. Pharmacotherapy offers promise for diabetes prevention, but with associated high costs, unacceptability to many patients, and potential toxicity. In this context, the potential role of chromium (Cr), an insulin co-factor, in IGT is of great interest. Chromium use is widespread, but evidence of any therapeutic effect is limited.

Proposed, therefore, is a randomized, double-blind, placebo controlled pilot trial conducted at the Yale Prevention Research Center, to investigate the effects of daily Cr for 6 months at two dose levels on serum measures of glucose tolerance, and on endothelial function, in adults with IGT, IFG, and IR. A modified crossover design will allow for paired and unpaired analyses including comparison of both 500 mcg and 1,000 mcg of Cr daily to placebo; comparison between 500 mcg and 1000 mcg of chromium; and evaluation of Cr washout time. The study is powered to detect a clinically meaningful effect of Cr supplementation at either dose on glucose control, and to compare the two doses for equivalence. The study will investigate effects of Cr on both measures of glucose tolerance (glucose, insulin, OGTT) and brachial artery endothelial function, thus combining serum measures with a physiologic test of Cr effects on the vasculature.

The proposed study will generate much needed data regarding the efficacy of Cr in those at risk for type II diabetes and offers the promise of guiding practice, as well as directing future study. By contributing to knowledge related to potential diabetes prevention strategies, this study addresses one of the more pressing public health issues in the US today. Risk to human subjects in this study is a minor increment over minimal due to the administration of nitroglycerin as a control in BARS testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* 18 years of age or older
* Identified to have impaired glucose tolerance (IGT), impaired fasting glucose (IFG), or insulin resistance.

According to the 1999 World Health Organization (WHO) report, IGT is diagnosed if the following two criteria are met: 1) Plasma glucose two hours after consuming 75g glucose (OGTT) is at least 7.8 mmol/l (140 mg/dl) but below 11.1 mmol/l (200 mg/dl) and 2) Fasting plasma glucose level is less than 7.0 mmol/l (126 mg/dl). IFG is diagnosed by a fasting plasma glucose concentration of 5.6 mmol/l (100 mg dl/l) or greater, but less than 7.0 mmol/l (126 mg dl/l). NCEP ATP III guidelines define 5 components of insulin resistance.

At least 3 of the 5 criteria are required for the diagnosis. These components are:

Abdominal obesity determined by waist circumference >102cm(>40in) in men or >88cm(>35in) in women; triglyceride level ≥150mg/dL; HDL-C <40mg/dL in men or <50mg/dL in women; blood pressure ≥ 130/≥85mm Hg; and fasting glucose ≥ 100mg/dL.

-Connecticut residents willing to travel to Griffin Hospital in Derby, CT

Exclusion Criteria:

* Known diabetes (Fasting Plasma Glucose > 126 mg/dl; 2-hour 75-g OGTT plasma glucose > 200 mg/dl;
* Diabetes diagnosed by a physician and confirmed by other clinical data);
* Self-reported hospitalization for treatment of heart disease in past 6 months;
* Impaired renal function as measured by labwork at initial screening (serum creatinine greater than 2.0 Serum creatinine and urine albumin excretion will be tested every six months throughout the study). Significant changes from baseline or to outside of threshold will be reported to the DSMB for appropriate action, including removal from the study.
* Self-reported pancreatitis. In the instance that potential subjects report that they are unsure whether they have been diagnosed with this condition, a primary medical doctor's note will be obtained confirming non-diagnosis before inclusion in the study.
* Self-reported recent or significant abdominal surgery;
* Self-reported pregnancy and/or intention become pregnancy during the study. Women of child-bearing age will consent to pregnancy testing at baseline, and will agree to avoiding pregnancy by reliable means throughout the duration of the study.
* Self-reported polycystic ovarian syndrome or irregular menses will be excluded from the study. (In the future, people with self-reported polycystic ovarian syndrome or irregular menses may be allowed in the study, however, because their conditions have the potential of affecting the outcome of BARS testing (a secondary outcome), they will be treated as a subset of the population during data analysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Serum Insulin | Baseline, 6, 12, 18 months
2-hour Oral Glucose Tolerance Test | Baseline, 6, 12, 18 months
Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) | Baseline, 6, 12, 18 months

SECONDARY OUTCOMES:
HbA1C | Baseline, 6, 12, 18 months
blood pressure | Baseline, 6, 12, 18 months
lipid profile (total cholesterol, LDL, HDL, TG) | Baseline, 6, 12, 18 months
BMI | Baseline, 6, 12, 18 months
urine albumin:creatinine ratio | Baseline, 6, 12, 18 months
endothelial function measures as percent flow-mediated dilitation (FMD). | Baseline, 6, 12, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David L Katz, MD, MPH, Principal Investigator — Yale University/Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

REFERENCES:
- [Result] Ali A, Ma Y, Reynolds J, Wise JP Sr, Inzucchi SE, Katz DL. Chromium effects on glucose tolerance and insulin sensitivity in persons at risk for diabetes mellitus. Endocr Pract. 2011 Jan-Feb;17(1):16-25. doi: 10.4158/EP10131.OR. PMID 20634174
- See also: Yale-Griffin Prevention Research Center — http://www.yalegriffinprc.org